CLINICAL TRIAL: NCT02474199
Title: Safety of Donor Alloantigen Reactive Tregs to Facilitate Minimization and/or Discontinuation of Immunosuppression in Adult Liver Transplant Recipients (CTOTC-12)
Brief Title: Donor Alloantigen Reactive Tregs (darTregs) for Calcineurin Inhibitor (CNI) Reduction
Acronym: ARTEMIS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation in Children (Other); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CTOTC-12
Record Dates: First submitted 2015-06-15; First posted 2015-06-17 (Estimated); Results first posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Liver Transplant Recipient; Living Donor (of the Respective Liver Transplant Recipient)
Keywords: Regulatory T Cells ( Treg); Donor Alloantigen Reactive Tregs (darTregs); Liver Transplant; Alloantigen Reactive Tregs; Calcineurin Inhibitors (CNI); immunosuppressants (IS)
MeSH Terms: interventions — Acetaminophen; Diphenhydramine; Immunosuppression Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- darTregs (Experimental): Donor Alloantigen Reactive Tregs (darTregs). Participants will receive a target dose of 400X10^6 darTregs (range 300-500 x10^6) infused intravenously (IV) over an approximate 20-30 minute interval
  Interventions: Biological: darTregs; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Immunosuppression (IS) Withdrawal; Procedure: Study Mandated Procedures

INTERVENTIONS:
Biological: darTregs — A single intravenous infusion as described administered over a 20-30 minute interval with close monitoring prior to, during, and after the infusion.
  Other Names: Donor Alloantigen Reactive Tregs
Drug: Acetaminophen — Pre-medication for darTregs infusion. A dose of 15 mg/kg will be administered 30 to 60 minutes prior to the darTregs infusion.
Drug: Diphenhydramine — Pre-medication for darTregs infusion. A dose of 1-2 mg/kg diphenhydramine will be administered 30 to 60 minutes prior to the darTregs infusion.
  Other Names: Diphenhydramine Hydrochloride
Drug: Immunosuppression (IS) Withdrawal — Subjects:1.) who fulfill study eligibility criteria will withdraw IS 2.) enter the study on calcineurin inhibitor (CNI) monotherapy or a CNI-based regimen with either Prednisone or MMF as a second IS medication 3.) will proceed with changes in CNI dosing according to the protocol's CNI withdrawal algorithm.During the last 2 weeks of IS withdrawal (e.g., Step 2 in algorithm -CNI reduced 25%-"pre darTregs"), a single dose of darTregs will be infused IV. The subject will then, if eligible, proceed with IS withdrawal within 2 weeks after the infusion. Eligible subjects meeting the primary endpoint of 75% reduction in CNI from baseline after darTregs will be offered the opportunity to continue IS withdrawal until complete discontinuation of IS.
  Other Names: IS Withdrawal; CNI based IS regimen
Procedure: Study Mandated Procedures — Blood draws (venipuncture); collection of peripheral blood mononuclear cells (PBMCs) by a procedure known as leukapheresis or venipuncture; buccal (cheek) swab for HLA typing; liver biopsies (per protocol and for cause).

SUMMARY:
This research study is for liver transplant recipients and their respective living donors.

The purpose of this study is:

1. To see if it is safe for liver recipients to receive one dose of donor reactive T regulatory cells (Tregs)
2. To see if the Tregs allows a liver recipient to take less, or completely stop medications normally taken after receiving an organ transplant.

DETAILED DESCRIPTION:
Doctors give drugs called immunosuppressants (IS) to people who receive a liver transplant. IS must be taken every day to prevent the body from injuring the transplanted liver by a process called rejection. Liver transplant recipients usually have to take these drugs for the rest of their lives. These drugs have harmful side effects. Researchers are looking for ways to keep a transplanted liver working normally with as little IS medications as possible. Finding a way to lower and then stop these medications will allow the liver recipient to avoid unwanted side effects.

Another area of research looks at how blood cells work to reject or accept an organ transplant. Studies show that some of the recipient's own cells, called T regulatory cells (Tregs), may play a part in accepting the transplanted liver and preventing rejection.

A recipient's Tregs can be grown in the laboratory to increase their number. Exposing the recipient's Tregs to the liver donor's cells will stimulate the Tregs that recognize the liver donor to grow vigorously. Giving these "donor reactive" Tregs back to the transplant recipient through a vein (intravenously) might allow a liver transplant recipient to take lower doses of IS, or perhaps to stop them altogether, without rejecting the liver.

The study team will collect information about the Treg infusion, liver tests and drug doses during IS withdrawal, and any problems that may arise in the study. Blood, liver tissue, and buccal (cheek) cells will be collected for research tests.

ELIGIBILITY:
Study Enrollment Inclusion Criteria:

* Subjects who meet all of the following criteria are eligible for enrollment:

  1. Able to understand and provide informed consent
  2. Have received a primary, solitary, living donor liver transplant more 24 months and less than 84 months ago
  3. Have a living donor who is willing to consent to a one time blood draw of 100 mLs to enable the manufacture of Donor Alloantigen Reactive Regulatory T cells (darTregs)
  4. Eighteen to 70 years of age at the time of study entry/consent
  5. Liver function test (LFT) results: have Alanine Aminotransferase (ALT)consistently <60 U/L and either alkaline phosphatase consistently <150 U/L or Gamma-glutamyl transferase (GGT) consistently <60 U/L
  6. Currently receiving a Calcineurin Inhibitor (CNI) with 12 hour trough levels consistently <6.0 ng/mL for tacrolimus; <150 ng/mL for cyclosporine
  7. Currently receiving CNI monotherapy or CNI and one of the following:

     1. Prednisone: maximum dose of 5mg daily
     2. Mycophenolate mofetil (MMF): maximum dose of 500 mg administered twice daily for Cellcept or 360mg twice daily for Myfortic.
  8. Female and male participants with reproductive potential must agree to use effective methods of birth control for the duration of the study.
  9. If history of Hepatocellular carcinoma (HCC), liver transplantation (LT) recipients who have:

     1. α-fetoprotein (AFP) less than 100 μg/L at the time of transplant AND
     2. Explanted liver:

        * with tumor burden within the Milan criteria and
        * without macro- or micro-vascular invasion and
        * without any lesions with poorly differentiated HCC and
        * without cholangiocarcinoma morphology
     3. Risk Estimation of Tumor Recurrence After Transplant (RETREAT) Score less than or equal to 3
  10. If history of HCC, at the time of enrollment, subjects must also:

      1. Be 36 months or more post-transplant AND
      2. Without evidence of recurrent HCC defined as:

         * AFP within normal limits for performing laboratory;
         * Confirmatory chest CT and
         * Confirmatory CT or MRI of the abdomen and pelvis.
  11. If history of hepatitis C virus (HCV) , recipients must be:

      1. Cured of HCV as defined by achieving Sustained virologic response (SVR) and be greater than or equal to six months after the end of treatment
      2. HCV RNA negative at time of study enrollment

Study Enrollment Exclusion Criteria:

* Participants who meet any of these criteria are not eligible for study enrollment:

  1. Transplant for liver disease secondary to autoimmune disease (e.g. autoimmune hepatitis, primary sclerosing cholangitis, or primary biliary cirrhosis)
  2. Matched at both human leukocyte antigen (HLA)-DR loci to the donor
  3. Organ, tissue or cell transplant prior to or after the primary solitary living donor liver transplant
  4. For subjects with hepatitis B, detectible hepatitis B virus (HBV) DNA
  5. History of malignancy within 5 years of enrollment. History of adequately treated in-situ cervical carcinoma and/or skin cancer (basal or squamous cell) will be permitted.
  6. Serologic evidence of human immunodeficiency 1 or 2 infection
  7. Epstein Barr Virus (EBV) seronegativity (EBV naïve) if living donor is EBV seropositive
  8. Cytomegalovirus (CMV) seronegativity (CMV naïve) if living donor is CMV seropositive
  9. Calculated Glomerular filtration rate (GFR) less than 50 mL/min/1.73m^2 at the time of enrollment
  10. An episode of Acute Rejection (AR) within one year of enrollment
  11. Systemic illness requiring or likely to require recurrent or chronic immunosuppression (IS) drug use
  12. Any chronic condition for which anti-coagulation cannot be safely interrupted for liver biopsy
  13. Positive pregnancy test
  14. Participation in any other studies that involved investigational drugs or regimens in the preceding year
  15. Any other condition, in the investigator's judgment, that increases the risk of darTregs infusion or prevents safe trial participation
  16. Unwilling or unable to adhere to study requirements and procedures
  17. Screening liver biopsy with any of the following histological criteria, as determined by the reading of a central pathologist.

darTregs Infusion Inclusion Criteria:

* Subjects must meet all criteria below to receive darTregs infusion:

  1. Stable liver tests, defined as ALT and either alkaline phosphatase or GGT either within normal limits OR <\=1.5 X baseline
  2. No detectible circulating EBV or CMV DNA prior to Treg infusion, assessed at the time of PBMC collection for manufacture
  3. For subjects with hepatitis B virus (HBV), no detectible circulating HBV DNA, assessed at the time of PBMC collection for manufacture
  4. Able to understand and provide informed consent.

darTregs Infusion Exclusion Criteria:

Subjects who meet any of these criteria are not eligible for darTregs infusion:

1. Diagnosis of AR after initiation of IS withdrawal
2. Any vaccination given within 28 days prior to Treg collection for Treg production
3. Receipt of a vaccination within 14 days prior to Treg infusion
4. Unacceptable darTregs product
5. Positive pregnancy test
6. Clinical evidence of viral syndrome less than 7 days prior to darTregs infusion.

Inclusion Criteria for Resuming IS Withdrawal after darTregs Infusion:

Subjects are eligible to resume IS withdrawal after darTregs infusion if all criteria below are met:

1. Subject received at least 100 x 10^6 darTregs
2. ALT and either alkaline phosphatase or GGT remain within normal limits or <\= 1.5 x baseline after darTregs infusion
3. For subjects with elevated liver tests as defined above, local pathology reading of liver biopsy 6-10 days after darTregs infusion is without AR according to Banff criteria
4. IS withdrawal resumes no later than 14 days after darTregs infusion
5. Site principal investigator determines it is acceptable for the study subject to resume IS withdrawal.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Feng, Principal Investigator — University of California at San Francisco; Jeffrey Bluestone, PhD, Study Chair — University of California at San Francisco; Qizhi Tang, PhD, Study Chair — University of California at San Francisco
Locations (3):
- United States (3):
  - University of California at San Francisco, San Francisco, California
  - Northwestern University Comprehensive Transplant Ctr, Chicago, Illinois
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Derived] Tang Q, Leung J, Peng Y, Sanchez-Fueyo A, Lozano JJ, Lam A, Lee K, Greenland JR, Hellerstein M, Fitch M, Li KW, Esensten JH, Putnam AL, Lares A, Nguyen V, Liu W, Bridges ND, Odim J, Demetris AJ, Levitsky J, Taner T, Feng S. Selective decrease of donor-reactive Tregs after liver transplantation limits Treg therapy for promoting allograft tolerance in humans. Sci Transl Med. 2022 Nov 2;14(669):eabo2628. doi: 10.1126/scitranslmed.abo2628. Epub 2022 Nov 2. PMID 36322627
- [Derived] Wood-Trageser MA, Lesniak D, Gambella A, Golnoski K, Feng S, Bucuvalas J, Sanchez-Fueyo A, Demetris AJ. Next-generation pathology detection of T cell-antigen-presenting cell immune synapses in human liver allografts. Hepatology. 2023 Feb 1;77(2):355-366. doi: 10.1002/hep.32666. Epub 2022 Aug 1. PMID 35819312
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Clinical Trials in Organ Transplantation in Children (CTOT-C) — https://www.ctotc.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between June 2016 and October 2018 at 3 clinical centers across the United States. A total of 15 participants were enrolled.
Pre-assignment Details: Five participants who signed informed consents did not proceed to immunosuppression withdrawal: 4 did not meet inclusion/exclusion criteria, 1 chose not to continue in the study.
Groups:
- Initiated Immunosuppression Withdrawal, Received darTregs: Initiated Immunosuppression Withdrawal, Received darTregs: Adult liver transplant recipients who signed informed consent, began immunosuppression withdrawal, and received the darTreg infusion. Adverse events were collected for these participants.
- Initiated Immunosuppression Withdrawal, Did Not Receive darTregs: Initiated Immunosuppression Withdrawal, Did Not Receive darTregs: Adult liver transplant recipients who signed informed consent, began immunosuppression withdrawal, and did not receive the darTreg infusion. Adverse events were collected for these participants.
- Did Not Initiate Withdrawal, Screening Biopsy Performed: Did Not Initiate Withdrawal, Screening Biopsy Performed: Adult liver transplant recipients who signed informed consent, had the protocol-mandated screening biopsy performed, and did not proceed to immunosuppression withdrawal. Adverse events were collected for these participants.
- Did Not Initiate Withdrawal, Screening Biopsy Not Performed: Did Not Initiate Withdrawal, Screening Biopsy Not Performed:
  Adult liver transplant recipients who signed informed consent, did not have the protocol-mandated screening biopsy performed, and did not proceed to immunosuppression withdrawal. Adverse events were not collected for these participants.
Period: Overall Study
Arm/Group | Initiated Immunosuppression Withdrawal, Received darTregs | Initiated Immunosuppression Withdrawal, Did Not Receive darTregs | Did Not Initiate Withdrawal, Screening Biopsy Performed | Did Not Initiate Withdrawal, Screening Biopsy Not Performed
Started | 5 | 5 (Insufficient numbers of darTregs for infusion (4 of these 5 participants)) | 2 | 3
Completed | 3 | 2 | 0 | 0
Not Completed | 2 | 3 | 2 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 1
Not completed — Did not receive Tregs due to insufficient manufacture | 0 | 1 | 0 | 0
Not completed — Did not meet eligibility criteria | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: All participants who initiated immunosuppression withdrawal. This population includes participants who received darTregs and participants who did not receive the darTregs infusion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Initiated Immunosuppression Withdrawal, Received darTregs | Initiated Immunosuppression Withdrawal, Did Not Receive darTregs | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (15.42) | 57.6 (19.03) | 53.2 (16.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10
Time Post-Transplant [Mean (Standard Deviation); unit: years] — This measure presents the time post-transplant at enrollment for all participants who initiated immunosuppression withdrawal (those who received darTregs and those who did not). Time is calculated for each participant as the number of years between their transplant date and their informed consent date.
  years | 3.3 (1.59) | 3.4 (1.43) | 3.4 (1.43)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Grade 3 or Higher Adverse Events (AEs) Deemed Attributable to darTreg Infusion
Description: The National Cancer Institute - Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 was used to grade the severity of all AEs. A participant was considered to have met this endpoint if they experienced at least one CTCAE Grade 3 or higher AE deemed attributable (i.e., considered at least possibly related) to darTreg infusion (infusion reaction, cytokine release syndrome).
Time Frame: From initiation of immunosuppression withdrawal to 24 weeks after darTregs infusion
Population: Participants who initiated immunosuppression withdrawal and received darTregs
Measure: Count of Participants; unit: Participants
Arm/Group | Initiated Immunosuppression Withdrawal, Received darTregs
Number analyzed (Participants) | 5
Participants | 0

2. Primary Outcome: Number of Participants With Study Defined Grade 3 or Higher Infections
Description: The following grading system was applied to AEs of infection:
  * Grade 1: asymptomatic; clinical or diagnostic observation only; intervention with oral antibiotic, antifungal, or antiviral agent only; no invasive intervention required
  * Grade 2: symptomatic; intervention with intravenous antibiotic, antifungal, or antiviral agent; invasive intervention may be required
  * Grade 3: any infection associated with hemodynamic compromise requiring pressors; any infection necessitating intensive care unit level of care; any infection necessitating operative intervention; any infection involving the central nervous system; any infection with a positive fungal blood culture; any proven or probable aspergillus infection; any tissue invasive fungal infection; any pneumocystis jiroveci infection
  * Grade 4: life-threatening infection
  * Grade 5: death resulting from infection
  A participant was considered to have met this endpoint if they experienced at least one Grade 3 or higher infection.
Time Frame: From initiation of immunosuppression withdrawal to 24 weeks after darTregs infusion
Population: All participants who initiated immunosuppression withdrawal. Since both groups initiated immunosuppression withdrawal, the participants who received darTregs were combined with the participants who did not receive the darTreg infusion to form the pre-defined group for assessment of this outcome.
Measure: Count of Participants; unit: Participants
Groups:
- Initiated Immunosuppression Withdrawal: All participants who initiated immunosuppression withdrawal. Since both groups initiated immunosuppression withdrawal, the participants who received darTregs were combined with the participants who did not receive the darTreg infusion to form the pre-defined group for assessment of this outcome.
Arm/Group | Initiated Immunosuppression Withdrawal
Number analyzed (Participants) | 10
Participants | 0

3. Primary Outcome: Number of Participants With Any Malignancy
Description: Number of participants with any malignancy, including Post -Transplant Lymphoproliferative Disorder (PTLD). PTLD is a specific type of malignancy that can occur following transplantation of a solid organ and is characterized by a proliferation of B cells, which may result in lymphoma.
Time Frame: From initiation of immunosuppression withdrawal to 24 weeks after darTregs infusion
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Initiated Immunosuppression Withdrawal
Number analyzed (Participants) | 10
Participants | 0

4. Primary Outcome: Proportion of Liver Transplant Recipients Who Are Able to Reduce Calcineurin Inhibitor Dosing by 75 Percent and Discontinue a Second Immunosuppression Drug (if Applicable) With Stable Liver Function Tests (LFTs) for ≥ 12 Weeks
Description: The ability to reduce baseline, standard of care calcineurin inhibitor dosing following transplantation was measured by determining the number of subjects who were able to tolerate a 75 percent reduction in their calcineurin inhibitors along with discontinuation of either prednisone or mycophenolate mofetil following initiation of immunosuppression withdrawal.
Time Frame: From initiation of immunosuppression withdrawal to 24 weeks after darTregs infusion
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Initiated Immunosuppression Withdrawal
Number analyzed (Participants) | 10
Proportion of Participants | 0.20 [0.0252 to 0.5561]

5. Secondary Outcome: Number of Liver Transplant Recipients Who Experience the Composite Outcome
Description: This measure includes refractory acute rejection, chronic rejection, re-transplantation, and death. Rejection was diagnosed based on local pathology. Participants are considered to have met this endpoint if they experience any one of these events at least once.
Time Frame: From initiation of immunosuppression withdrawal to 52 weeks after darTreg infusion
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Initiated Immunosuppression Withdrawal
Number analyzed (Participants) | 10
Participants | 0

6. Secondary Outcome: Number of Participants Who Experience at Least One Episode of Biopsy Proven Acute Rejection, Clinical Acute Rejection, or Chronic Rejection
Description: A participant was considered to have met this endpoint if they experienced at least one episode of biopsy proven acute rejection, clinical acute rejection, or chronic rejection based on local pathology.
  Biopsy proven acute rejection was assessed as Grade I or higher based on the Banff (1997) global criteria featuring the following grades:
  * Indeterminate
  * Grade I Mild Acute Rejection
  * Grade II Moderate Acute Rejection
  * Grade III Severe Acute Rejection.
  Clinical AR was determined based on the participant receiving treatment for rejection with or without biopsy confirmation of rejection.
  Chronic rejection was determined by the presence of abnormal total and direct bilirubin in the conjunction with liver pathology fulfilling the Banff (2000) criteria as outlined:
  * Early Stage Chronic Rejection
  * Late Stage Chronic Rejection.
Time Frame: From initiation of immunosuppression withdrawal to 52 weeks after darTreg infusion
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Initiated Immunosuppression Withdrawal
Number analyzed (Participants) | 10
Participants | 5

7. Secondary Outcome: Count of Participants by Severity of Biopsy Proven Acute Rejection and/or Chronic Rejection
Description: Participants are counted in each grade of rejection they experienced; however, a participant is only counted once within a specific grade. Biopsy proven acute rejection and Chronic rejection were graded based on local pathology according to the Banff (1997 for Acute Rejection; 2000 for Chronic Rejection) global assessment criteria as outlined below.
  Biopsy proven acute rejection was assessed as Grade I or higher using the following grades:
  * Indeterminate
  * Grade I Mild Acute Rejection
  * Grade II Moderate Acute Rejection
  * Grade III Severe Acute Rejection.
  Chronic rejection was determined by the presence of abnormal total and direct bilirubin in the conjunction with liver pathology fulfilling the Banff criteria as outlined:
  * Early Stage Chronic Rejection
  * Late Stage Chronic Rejection.
Time Frame: From initiation of immunosuppression withdrawal to 52 weeks after darTregs infusion
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Initiated Immunosuppression Withdrawal
Number analyzed (Participants) | 10
Participants
  Mild Acute Rejection | 2
  Moderate Acute Rejection | 0
  Severe Acute Rejection | 0
  Early Stage Chronic Rejection | 0
  Late Stage Chronic Rejection | 0

8. Secondary Outcome: Number of Participants Achieving Efficacy Status Post Receipt of a Single Intravenous (IV) Dose of Donor Alloantigen Reactive Regulatory T Cells (darTregs)
Description: Efficacy was assessed by determining the number (and percentage) of participants who have received darTreg infusion and are identified as operationally tolerant, defined by maintaining stable allograft function (assessed by liver tests) and histology (determined by central pathologist reading in comparison to screening liver biopsy at study entry) in the absence of immunosuppression for one year.
Time Frame: From initiation of immunosuppression withdrawal to 52 weeks after darTreg infusion
Population: Participants who initiated immunosuppression withdrawal and received darTregs.
Measure: Count of Participants; unit: Participants
Arm/Group | Initiated Immunosuppression Withdrawal, Received darTregs
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years (24 months)
Description: Only adverse events (AEs) grade 2 or higher were collected. Only AEs associated with protocol mandated liver biopsy were collected from the time of the biopsy to the initiation of initial immunosuppression (IS) withdrawal. All SAEs, regardless of relationship or expectedness to blood draw or liver biopsy with research specimen collection, IS withdrawal, or Treg infusion were to be reported within 24 hours of awareness.
Arm/Group | Initiated Immunosuppression Withdrawal, Received darTregs | Initiated Immunosuppression Withdrawal, Did Not Receive darTregs | Did Not Initiate Withdrawal, Screening Biopsy Performed
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 4/5 | 1/5 | 0/2
Other Adverse Events (participants affected / at risk) | 0/5 | 2/5 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initiated Immunosuppression Withdrawal, Received darTregs (N=5) | Initiated Immunosuppression Withdrawal, Did Not Receive darTregs (N=5) | Did Not Initiate Withdrawal, Screening Biopsy Performed (N=2)
Transplant rejection (Immune system disorders) | 4 (4) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initiated Immunosuppression Withdrawal, Received darTregs (N=5) | Initiated Immunosuppression Withdrawal, Did Not Receive darTregs (N=5) | Did Not Initiate Withdrawal, Screening Biopsy Performed (N=2)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT02474199/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT02474199/SAP_001.pdf